CLINICAL TRIAL: NCT04176042
Title: Community-Level Daytime Sleepiness: Social-Environmental Determinants, Consequences, and Impact of Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Michael A. Grandner, Associate Professor of Psychiatry, Psychology, and Medicine; Director, Sleep & Health Research Program, University of Arizona, University of Arizona
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1906742940
Record Dates: First submitted 2019-11-08; First posted 2019-11-25 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Daytime Sleepiness
Keywords: Daytime Sleepiness; Environmental Determinants; Sleep Beliefs; Sleep Attitudes; Educational Intervention; Focus Group; Epworth Sleepiness Scale
MeSH Terms: conditions — Disorders of Excessive Somnolence

STUDY DESIGN:
Intervention Model Description: 4-WEEK TRACKS All 28 participants will be randomized to one of two 4-week tracks (N=14 each). The study design (crossover) dictates that all participants must complete a questionnaire at identical time points; therefore, participants in track 2 will perform a baseline questionnaire at the same time as track 1 participants perform a baseline questionnaire for their intervention. Also, participants in track 1 will complete the follow up at the same time as track 2 participants perform a baseline questionnaire for their intervention.
Who Masked: Participant
Masking Description: All 28 participants will be randomized to one of two 4-week tracks (N=14 each).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Track 1 (Experimental): Subjects will be randomized to one of two 4-week tracks.
  Track 1 (intervention + follow-up) will consist of the following:
  Subjects will be randomized to one of two 4-week tracks. Track 1 (intervention + follow-up) will consist of the following: Prior to the session, within 72 hours of the scheduled 2-hour education invention participants will complete a baseline questionnaire battery consisting of measures including demographics, medical history and sleep. After completion, a 2-hour educational presentation will take place with a question-and-answer session. Participants will then complete post-intervention questionnaires to assess immediate impact of the session on knowledge, beliefs and practices. After 4 weeks, Track 1 participants will be contacted and will be asked to re-complete all baseline questionnaires (see above), in order to evaluate changes over 4 weeks.
  Interventions: Behavioral: Track 1
- Track 2 (Active Comparator): Subjects will be randomized to one of two 4-week tracks. Track 2 (wait list + intervention) will consist of the following: Prior to the session, within 72 hours of the scheduled 2-hour education invention for Track 1 participants will complete the same baseline questionnaire battery.
  An identical intervention session, scheduled 4 weeks into the future. At that time, an identical procedure to the other track will be followed, including the pretest questionnaires, 2-hour session, and post-session assessment. No additional 4-week follow-up will be performed.
  Interventions: Behavioral: Track 2

INTERVENTIONS:
Behavioral: Track 1 — Intervention + Follow-up
  Arms: Track 1
Behavioral: Track 2 — Wait list + Intervention
  Arms: Track 2

SUMMARY:
The purpose of this study is to examine daytime sleepiness in a community context. This includes examining sleepiness in a large sample in terms of social/behavioral/environmental predictors and health-related outcomes, as well as examining the role of a sleep education intervention in a smaller sample for promoting healthy beliefs/attitudes about sleepiness.

DETAILED DESCRIPTION:
Increasing attention has focused on the role of sleep in public health. Approximately 1/3 of Americans sleep ≤6h per night, an amount that has been deemed sub-optimal by the American Academy of Sleep Medicine and Sleep Research Society, the National Sleep Foundation, American Thoracic Society, and the American Heart Association. These consensus statements echo findings from many reviews on this topic. This is alarming, given epidemiologic and experimental research showing that reduced sleep time is associated with a variety of negative health outcomes including obesity, diabetes, cardiovascular disease, and mortality. As such, short sleep represents an unmet public health problem. The community-level daytime impacts of insufficient sleep are still not well characterized, though.

Previous studies have associated habitual short sleep duration with important adverse cardiometabolic outcomes, including weight gain, obesity, diabetes, cardiovascular disease, stress, etc. They suggest that those that report short sleep may be more likely to experience functional impairments and are less likely to engage in behaviors consistent with a healthy lifestyle. A proposed mechanism of these relationships is that insufficient sleep duration triggers metabolic disturbances and increased immune response, resulting in appetite dysregulation, adverse cardiovascular outcomes, and resultant disease states. In addition to cardiometabolic effects, behavioral and functional consequences of short sleep have been well-documented. For example, short sleepers are more likely to exhibit difficulties initiating and/or maintaining sleep, daytime sleepiness, drowsy driving, and other impairments as a result of sleep loss. Laboratory studies have extensively documented neurocognitive and behavioral effects of sleep loss, including increased objective sleepiness, impaired vigilance using computer-based psychomotor assessments, and deficits in working memory, decision-making, and executive function, as assessed using standardized neuropsychologic and neuroimaging techniques. Although much of the focus on sleep as a public health issue has been on insufficient sleep at night, relatively little has focused on the role of daytime sleepiness. The investigator's previous work has shown that the prevalence of daytime tiredness is approximately 18-19% among working-age adults in the US. This is in line with other studies, which have estimated the population burden of excessive daytime sleepiness to be between 10-25%. Daytime sleepiness is a well-documented result of sleep deprivation, but it can also be a result of sleep apnea, sleep fragmentation, and other causes. The role of daytime sleepiness as an important dimension of sleep that impacts public health has not been sufficiently explored. The present study aims to examine daytime sleepiness in a large community sample in terms of social/behavioral/environmental predictors and health-related outcomes.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study trial, subjects must:

* Subject is a male or female, 20-60 years of age, inclusive.
* Subject is not pregnant.
* Subject obtains a score of >10 on the Epworth Sleepiness Scale, indicating high daytime sleepiness.
* Subject presents no apparent unstable and/or major medical or psychiatric conditions that may contribute to sleepiness.
* Subject is fluent in English.
* Subject is willing to take part in this study.

Exclusion Criteria:

* Subject is under the age of 20 or over the age of 60.
* Subject is pregnant.
* Subject presents apparent unstable and/or major medical or psychiatric conditions that may contribute to sleepiness.
* Subject is not fluent in English.
* Subject obtained a score of <10 on the Epworth Sleepiness Scale.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change of Epworth Sleepiness Scale (ESS) score across specific time points for Track 1 | Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to follow up (after 4 weeks).
  ESS is a standard measure to assess daytime sleepiness and consists of 8 items ranging from "No chance of dozing" to "High chance of dozing" that evaluate sleep propensity in a range of situations.
Change of Epworth Sleepiness Scale (ESS) score across specific time points for Track 2 | Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to pre-intervention (after 4 weeks).
  ESS is a standard measure to assess daytime sleepiness and consists of 8 items ranging from "No chance of dozing" to "High chance of dozing" that evaluate sleep propensity in a range of situations.
Changes in Sleep Practices and Attitudes Questionnaire (SPAQ) score for Track 1 | Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to immediately post-intervention (2 hours), and to follow up (after 4 weeks)
  This questionnaire assesses habitual sleep behaviors associated with sleep and potential sleep problems.
Changes in Sleep Practices and Attitudes Questionnaire (SPAQ) score for Track 2 | Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to pre-intervention (after 4 weeks), and to immediately post-intervention (2 hours)
  This questionnaire assesses habitual sleep behaviors associated with sleep and potential sleep problems.
Changes in Sleep Beliefs Scale (SBS) score for Track 1 | Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to immediately post-intervention (2 hours), and to follow up (after 4 weeks)
  The SBS is a revised version of the Sleep Hygiene Awareness and Practice Scale. Possessing a simplified scoring method, the SBS consists of the nine most salient questions from the previous scale, along with 11 relevant additions. The scale requires respondents to indicate how certain behaviors (e.g., drug consumption, daytime and evening activities) can influence the quality and quantity of an individual's sleep, with answers ranging from "positive effect" (on sleep) to "negative effect" (on sleep).
Changes in Sleep Beliefs Scale (SBS) score for Track 2 | Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to pre-intervention (after 4 weeks), and to immediately post-intervention (2 hours)
  The SBS is a revised version of the Sleep Hygiene Awareness and Practice Scale. Possessing a simplified scoring method, the SBS consists of the nine most salient questions from the previous scale, along with 11 relevant additions. The scale requires respondents to indicate how certain behaviors (e.g., drug consumption, daytime and evening activities) can influence the quality and quantity of an individual's sleep, with answers ranging from "positive effect" (on sleep) to "negative effect" (on sleep).
Changes in Dysfunctional Beliefs About Sleep Scale score for Track 1 | Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to immediately post-intervention (2 hours), and to follow up (after 4 weeks)
  Consisting of 28 items, the scale evaluates sleep-related beliefs, querying respondents' expectations and attitudes regarding the causes, consequences, and potential treatments of sleep issues, with answers ranging from 0-"Strongly Disagree" to 10-"Strongly Agree".
Changes in Dysfunctional Beliefs About Sleep Scale score for Track 2 | Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to pre-intervention (after 4 weeks), and to immediately post-intervention (2 hours)
  Consisting of 28 items, the scale evaluates sleep-related beliefs, querying respondents' expectations and attitudes regarding the causes, consequences, and potential treatments of sleep issues, with answers ranging from 0-"Strongly Disagree" to 10-"Strongly Agree".

SECONDARY OUTCOMES:
Qualitative Themes in Sleep Beliefs (Discussed in a group setting) | Focus Group [Day 0]
  Focus Group to gather qualitative themes guided by the following questions:
  1. What is healthy sleep?
  2. What is unhealthy sleep?
  3. What is sleepiness?
  4. How does sleepiness affect you?
  5. What is the most important thing about your sleepiness?
  6. What do you do about your sleepiness?
Demographics and Personal Information | Track 1: Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to follow up (after 4 weeks). Track 2: Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to pre-intervention (after 4 weeks).
  This measure includes questions about age, sex, education level, relationship status, employment, status, and race/ethnicity.
Medical History | Track 1: Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to follow up (after 4 weeks). Track 2: Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to pre-intervention (after 4 weeks).
  Self-report questions about medical history, including family medical history
Fatigue Severity Scale (FSS) | Track 1: Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to follow up (after 4 weeks). Track 2: Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to pre-intervention (after 4 weeks).
  FSS is a well-validated 9-item clinical measure that assesses overall levels of mental and physical fatigue, with answers ranging from 1- "Strongly Disagree" to 7-"Strongly Agree".
Sleep Timing Questionnaire (STQ) | Track 1: Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to follow up (after 4 weeks). Track 2: Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to pre-intervention (after 4 weeks).
  STQ assesses weekday and weekend sleep timing and sleep duration, as well as variability in sleep timing, with responses in the form of # of minutes (i.e. 25 minutes) or hourly times (i.e. 7:00 pm).
Insomnia Severity Index (ISI) | Track 1: Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to follow up (after 4 weeks). Track 2: Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to pre-intervention (after 4 weeks).
  ISI is a brief (7-item) insomnia screening tool that is the gold standard for quantifying severity of clinical insomnia symptoms.
Sleep Disorders Symptom Check List | Track 1: Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to follow up (after 4 weeks). Track 2: Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to pre-intervention (after 4 weeks).
  a 20 question instrument was developed to screen for six sleep disorders (insomnia, obstructive sleep apnea, restless legs syndrome/periodic limb movement disorder, circadian rhythm sleep-wake disorders, narcolepsy, and parasomnias) and evaluated psychometrically. Answers range from "Never" to ">5 times a week" .
Patient Health Questionnaire (PHQ9) | Track 1: Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to follow up (after 4 weeks). Track 2: Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to pre-intervention (after 4 weeks).
  The PHQ9 will screen for depression symptoms. It is a multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression: It incorporates DSM-IV depression diagnostic criteria with other leading major depressive symptoms into a brief self-report tool. Participants with a score >9 will be excluded. A total score is calculated for this tool.
Generalized Anxiety Disorder 7- Item Scale (GAD-7) | Track 1: Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to follow up (after 4 weeks). Track 2: Changes from Baseline (approximately 7 days after Focus Group [Day 0]) to pre-intervention (after 4 weeks).
  is a self-reported questionnaire for screening and severity measuring of generalized anxiety disorder. It contains 7 items with answers ranging from "Not at all" to "Nearly every day".

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Grandner, PhD, MTR, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Department of Psychiatry Research Facilities, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No